CLINICAL TRIAL: NCT06573931
Title: Lumbar Erector Spinae Plane Block vs Fascia Iliaca Block vs Lumbar Plexus Block for Postoperative Analgesia for Total Hip Arthroplasty: A Randomized Clinical Trial
Brief Title: Lumbar Erector Spinae Plane Block vs Fascia Iliaca Block vs Lumbar Plexus Block for Postoperative Analgesia for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR760/7/24
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Erector Spinae Plane Block; Fascia Iliaca Block; Lumbar Plexus Block; Analgesia; Total Hip Arthroplasty
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbar Erector Spinae Plane Block (Experimental): Patients will receive lumbar erector spinae plane block at the end of surgery.
  Interventions: Other: Lumbar Erector Spinae Plane Block
- Fascia Iliaca Block (Experimental): Patients will receive fascia iliaca block at the end of surgery.
  Interventions: Other: Fascia Iliaca Block
- Lumbar Plexus Block (Experimental): Patients will receive lumbar plexus block at the end of surgery.
  Interventions: Other: Lumbar Plexus Block

INTERVENTIONS:
Other: Lumbar Erector Spinae Plane Block — Patients will receive lumbar erector spinae plane block at the end of surgery.
  Arms: Lumbar Erector Spinae Plane Block
Other: Fascia Iliaca Block — Patients will receive fascia iliaca block at the end of surgery.
  Arms: Fascia Iliaca Block
Other: Lumbar Plexus Block — Patients will receive lumbar plexus block at the end of surgery.
  Arms: Lumbar Plexus Block

SUMMARY:
This study aims to compare lumbar erector spinae plane block, fascia iliaca block, and lumbar plexus block for postoperative analgesia for hip surgery.

DETAILED DESCRIPTION:
Approximately 500,000 hip arthroplasties are performed each year in the United States. Traditionally, this procedure has been performed under general anesthesia. However, neuraxial and regional anesthesia have become more commonly utilized to aid in postoperative analgesia and reduce the side effects of opioids, namely sedation, nausea, and vomiting. Postoperative pain control has a significant impact on earlier ambulation, initiation of physical therapy, better functional recovery, and overall patient satisfaction.

Lumbar erector spinae plane block (LESPB) was reported to lead to effective postoperative analgesia in hip and proximal femoral surgery.

The fascia iliaca block (FIB) is an established and effective technique, especially when US guidance and proximal approaches are used.

lumbar plexus block (LPB) could be safe because of the targeted somatic nerve block in the psoas region which prevents dispensable sympathetic block even in cardiovascular-compromised patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Undergoing total hip arthroplasty under spinal anesthesia.

Exclusion Criteria:

* Obesity (Body Mass Index > 30 kg/m2).
* Allergy to any drug used in the study.
* Contraindications to spinal anesthesia (such as Thrombocytopenia (platelets <100,000/mCL) and coagulopathy (INR >1.4 or insufficient time since stopping systemic anticoagulation)).
* Epilepsy.
* Psychiatric disease.
* Pre-existing neurologic deficits or neuropathies.
* Pregnancy.
* Pre-existing alcohol/opioid use disorder.
* Previously diagnosed with chronic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of block to first dose of morphine administrated) will be recorded.

SECONDARY OUTCOMES:
Total morphine consumption in the 1st 24h | 24 hours postoperatively
  Rescue analgesia will be provided by patient-controlled analgesia (PCA) with intravenous morphine (no basal rate; bolus 1 mg, lockout 10 minutes, maximum dose 20 mg in 4 h), which will be started if the numeric rating scale (NRS)> 3. NRS will be assessed at PACU, 4, 8, 16, and 24 h postoperatively.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at PACU, 4, 8, 16, and 24 h postoperatively.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as Bradycardia, hypotension, postoperative nausea and vomiting (PONV), or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.